CLINICAL TRIAL: NCT03621865
Title: A Comparative Pharmacokinetic Study in Healthy Volunteers to Evaluate the Ability of TURMIPURE GOLD Formulation to Enhance the Bioavailability of Curcuminoids
Brief Title: A Comparative Pharmacokinetic Study to Evaluate the Ability of a New Formulation to Enhance Curcuminoids Bioavailability
Acronym: TURBIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Givaudan France Naturals (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2018_A01390-55
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: bioavailability; pharmacokinetic study; curcuminoids; curcumin; healthy volunteers
MeSH Terms: interventions — tetraethylpyrazine

STUDY DESIGN:
Intervention Model Description: This pharmacokinectic study is designed as a monocentric, randomized, cross-over, pilot and open clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- subject sequence 1 (Experimental): subject allocation sequence 1. Intervention: The subject will receive the five products (TG, STE, NOV, PHYT or TEP) in a certain order.
  Interventions: Dietary Supplement: TG; Dietary Supplement: STE; Dietary Supplement: NOV; Dietary Supplement: PHYT; Dietary Supplement: TEP
- subject sequence 2 (Experimental): subject allocation sequence 2. IIntervention: The subject will receive the five products (TG, STE, NOV, PHYT or TEP) in a certain order.
  Interventions: Dietary Supplement: TG; Dietary Supplement: STE; Dietary Supplement: NOV; Dietary Supplement: PHYT; Dietary Supplement: TEP
- subject sequence 3 (Experimental): subject allocation sequence 3. Intervention: The subject will receive the five products (TG, STE, NOV, PHYT or TEP) in a certain order.
  Interventions: Dietary Supplement: TG; Dietary Supplement: STE; Dietary Supplement: NOV; Dietary Supplement: PHYT; Dietary Supplement: TEP
- subject sequence 4 (Experimental): subject allocation sequence 4. Intervention: The subject will receive the five products (TG, STE, NOV, PHYT or TEP) in a certain order.
  Interventions: Dietary Supplement: TG; Dietary Supplement: STE; Dietary Supplement: NOV; Dietary Supplement: PHYT; Dietary Supplement: TEP
- subject sequence 5 (Experimental): subject allocation sequence 5. Intervention: The subject will receive the five products (TG, STE, NOV, PHYT or TEP) in a certain order.
  Interventions: Dietary Supplement: TG; Dietary Supplement: STE; Dietary Supplement: NOV; Dietary Supplement: PHYT; Dietary Supplement: TEP
- subject sequence 6 (Experimental): subject allocation sequence 6. Intervention: The subject will receive the five products (TG, STE, NOV, PHYT or TEP) in a certain order.
  Interventions: Dietary Supplement: TG; Dietary Supplement: STE; Dietary Supplement: NOV; Dietary Supplement: PHYT; Dietary Supplement: TEP
- subject sequence 7 (Experimental): subject allocation sequence 7. Intervention: The subject will receive the five products (TG, STE, NOV, PHYT or TEP) in a certain order.
  Interventions: Dietary Supplement: TG; Dietary Supplement: STE; Dietary Supplement: NOV; Dietary Supplement: PHYT; Dietary Supplement: TEP
- subject sequence 8 (Experimental): subject allocation sequence 8. Intervention: The subject will receive the five products (TG, STE, NOV, PHYT or TEP) in a certain order.
  Interventions: Dietary Supplement: TG; Dietary Supplement: STE; Dietary Supplement: NOV; Dietary Supplement: PHYT; Dietary Supplement: TEP
- subject sequence 9 (Experimental): subject allocation sequence 9. Intervention: The subject will receive the five products (TG, STE, NOV, PHYT or TEP) in a certain order.
  Interventions: Dietary Supplement: TG; Dietary Supplement: STE; Dietary Supplement: NOV; Dietary Supplement: PHYT; Dietary Supplement: TEP
- subject sequence 10 (Experimental): subject allocation sequence 10. Intervention: The subject will receive the five products (TG, STE, NOV, PHYT or TEP) in a certain order.
  Interventions: Dietary Supplement: TG; Dietary Supplement: STE; Dietary Supplement: NOV; Dietary Supplement: PHYT; Dietary Supplement: TEP

INTERVENTIONS:
Dietary Supplement: TG — Turmipure GOLD™ 30% curcuminoids (300 mg)
  Other Names: Turmipure GOLD™
Dietary Supplement: STE — Standard turmeric powder extract 95% curcuminoids (1500 mg)
  Other Names: Standard turmeric powder extract
Dietary Supplement: NOV — Novasol® Liquid micellar formulation 6% curcuminoids (1000 mg)
Dietary Supplement: PHYT — Meriva® Turmeric Phytosome formulation 20% curcuminoids (1000 mg)
Dietary Supplement: TEP — Turmeric extract C3 complex® 95% curcuminoids (1500mg) + BioPerine® 95% piperine (15 mg)

SUMMARY:
The rhizome of Curcuma longa (turmeric) is commonly used as a spice and for its medicinal properties traditionally in Asian countries. Turmeric extract usually contains 95% curcuminoids with a specific ratio (approximately 75-80% curcumin, 15-20% demethoxycurcumin (DMC), and 0-10% bisdemethoxycurcumin (BDMC)).

Curcuminoids have higher solubility in organic solvents than in water. As a consequence, curcuminoids have low aqueous solubility and poor gastrointestinal absorption. They also exhibit rapid metabolism and systemic elimination and are therefore known to have limited bioavailability, which limits the use of turmeric extract in general health care and as an adjunct in managing various diseases. In order to improve the bioavailability of curcumin, several approaches have been undertaken. The use of adjuvant like piperine that interferes with glucuronidation; liposomal curcumin, nanoparticles, phospholipid complex; and structural analogues of curcumin.

Recently, Naturex has developed a dried emulsion formulation using a turmeric extract mixed together with a quillaja extract, sunflower oil and arabic gum. This formulation is highly dispersible in water and should therefore improve the bioavailability of curcuminoids. The aim of this study is to assess the bioavailability of curcuminoids and their metabolites after oral intake of 4 turmeric extract-based formulations in comparison to a standard unformulated turmeric extract.

DETAILED DESCRIPTION:
The rhizome of Curcuma longa (turmeric) is commonly used as a spice and for its medicinal proprieties traditionally in Asian countries. Turmeric has been studying in different therapeutic areas. Antioxidant, anti-inflammatory (respiratory system, joints and digestive), antimutagenic, antimicrobial, neurological disease, hepatoprotective and anticancer properties are supported by in vitro and in vivo data.

Curcumin has been studied as the main bioactive component of turmeric associated to its potential health effect. However, besides curcumin, others components have been identified (demethoxycurcumin DMC and bisdemethoxycurcumin BDMC); this group of coumpounds are named together "curcuminoids". Curcuminoids are natural yellow-orange pigments and hydrophobic polyphenols derived from the rhizome of the herb Curcuma longa. They are commonly isolated from the spice and food-coloring agent turmeric. Extracts of turmeric generally contain 75-80% curcumin, 15-20% DMC, and 0-10% BDMC. Regarding the intrinsic property, curcuminoids have higher solubility in organic solvents than in water. As a consequence, curcuminoids have low aqueous solubility and poor gastrointestinal absorption. They also exhibit rapid metabolism and systemic elimination.

This leads to the conclusion that curcuminoids from turmeric extract have low bioavailability, which limits its use in general health care and as an adjunct in managing various diseases. In order to improve the bioavailability of curcumin, several approaches have been undertaken. The use of adjuvant like piperine that interferes with glucuronidation; liposomal curcumin, nanoparticles, phospholipid complex; and structural analogues of curcumin.

Recently, Naturex has developed a dried emulsion formulation using a turmeric extract mixed together with a quillaja extract, sunflower oil and arabic gum. This formulation is highly dispersible in water and should therefore improve the bioavailability of curcuminoids. The aim of this study is to assess the bioavailability of curcuminoids and their metabolites after oral intake of 4 turmeric extract-based formulations in comparison to a standard unformulated turmeric extract.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years (limits included),
* BMI between 19 and 25 kg/m² (limits included),
* Weight stable within ±3kg in the last three months,
* With routine blood chemistry values within the normal range
* For women: Non menopausal with the same reliable contraception since at least 3 cycles before the beginning of the study and agreeing to keep it during the entire duration of the study (condom with spermicidal gel and estrogen/progestin combination contraception accepted) or menopausal without or with hormone replacement therapy (estrogenic replacement therapy begun from less than 3 months excluded),
* Non smoking or with tobacco consumption ≤ 5 cigarettes / day and agreeing not to smoke during all experimental sessions (V1 to V5),
* Agreeing not to consume food, drink and condiment containing curcumin, turmeric (curcuma longa Linn.) or curry for 1 week prior to and throughout the entire study,
* Good general and mental health with in the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination,
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form,
* Affiliated with a social security scheme,
* Agreeing to be registered on the volunteers in biomedical research file

Exclusion Criteria:

* Suffering from a metabolic or endocrine disorder such as diabetes, uncontrolled or controlled thyroidal trouble or other metabolic disorder,
* Suffering from a severe chronic disease (e.g. cancer, HIV, renal failure, ongoing hepatic or biliary disorders, chronic inflammatory digestive disease, arthritis or other chronic respiratory trouble, etc.) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator (e.g. celiac disease),
* Suffering from liver diseases
* Current disease states that are contraindicated to subjects with dietary supplementation: chronic diarrhea, constipation or abdominal pain, Inflammatory bowel diseases (Crohn's disease or ulcerative colitis), Cirrhosis, chronic laxatives use…,
* Suffering from Irritable Bowel Syndrome (IBS) diagnosed by a medical doctor and treated with chronic medication,
* Having medical history of current pathology which could affect the study results or expose the subject to an additional risk according to the investigator,
* Recent gastroenteritis or food borne illness such as confirmed food poisoning (less than 1 month),
* Who made a blood donation in the 3 months before the V0 visit or intending to make it within 3 months ahead,
* With a low venous capital not allowing to perform kinetic of blood samples according to the investigator's opinion,
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient and/or of the standard meals (gluten intolerance, celiac disease, etc….)
* Pregnant or lactating women or intending to become pregnant within 3 months ahead,
* Exhibiting alcohol or drug dependence
* On any chronic drug treatment (for example anticoagulant, antihypertensive treatment, treatment thyroid, asthma treatment, anxiolytic, antidepressant, lipid-lowering treatment, corticosteroids, phlebotonic, veino-tonic, drug with impact on blood circulation …) excepting oral and local contraceptives,
* Currently taking (and during the past 3 months) any supplementation from botanical origins
* Having consumed curcumin-containing food supplements (curcumin, turmeric and curry) or foods (curcumin, turmeric, E100, and curry) defined as at least 3 times per week and for 2 weeks prior to testing
* Currently taking (and during the past 3 months) any prebiotics or probiotics supplementation from food or from dietary supplements
* With significant change in food habits or in physical activity in the 3 months before the V0 visit or not agreeing to keep them unchanged throughout the study,
* Trying to lose weight with a current or planned in the next 3 months specific diet (hyper or hypocaloric, vegan, vegetarian…) or exercice regimen
* With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator,
* Consuming more than 3 standard drinks of alcoholic beverage daily for men or 2 daily for women or not agreeing to keep his alcohol consumption habits unchanged throughout the study,
* Having a lifestyle deemed incompatible with the study according to the investigator including high level physical activity (defined as more than 10 hours of significant physical activity a week, walking excluded),
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial,
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros,
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision,
* Presenting a psychological or linguistic incapability to sign the informed consent,
* Impossible to contact in case of emergency.

After V0 biological analyses the subject will be considered as non-eligible to the study on the following criteria:

- Control record (Glycaemia, GGT, ASAT, ALAT, Urea, Creatinine and Complete blood count) with clinically significant abnormality according to the investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Dose-normalized AUC of total curcuminoids plasmatic concentration | from 0 to 24 hours
  The primary endpoint is the dose-normalized AUC of total curcuminoids (sum of curcumin, DMC, BDMC and their metabolites) plasmatic concentration from 0 to 24 hours (AUC0-24h/dose) (expressed in µg.h/mL/mg). The dose-normalized AUC is the AUC normalized to curcuminoids intake by dividing the observed AUC by the corresponding curcuminoids dosage of each administration The following time-points are considered: T0, T15, T30, T45, T60, T90, T120, T240, T60, T480, T24H. T-10 will be considered as baseline value (T0) for AUC calculation. The primary comparison is Turmipure Gold 300 mg vs Standard turmeric 1500 mg powder extract.

SECONDARY OUTCOMES:
AUC of total curcuminoids plasmatic concentration | from 0 to 24 hours
  AUC of total curcuminoids plasmatic concentration from 0 to 24 hours (AUC0-24h, expressed in µg.h/mL);
AUC of curcuminoids separately (curcumin, DMC, BDMC) plasmatic concentrations | from 0 to 24 hours
  AUC of curcuminoids separately (curcumin, DMC, BDMC) plasmatic concentrations from 0 to 24 hours (AUC0-24h, expressed in µg.h/mL);
AUC of curcuminoids metabolites plasmatic concentrations | from 0 to 24 hours
  AUC of curcuminoids metabolites plasmatic concentrations from 0 to 24 hours (AUC0-24h, expressed in µg.h/mL);
AUC of total curcuminoids plasmatic concentration normalized to curcuminoids intake | from 0 to 8 hours
  AUC of total curcuminoids plasmatic concentration from 0 to 8 hours normalized to curcuminoids intake (AUC0-8h/dose, expressed in µg.h/mL/mg);
AUC of total curcuminoids plasmatic concentration | from 0 to 8 hours
  AUC of total curcuminoids plasmatic concentration from 0 to 8 hours (AUC0-8h) (expressed in µg.h/mL);
AUC of curcuminoids separately (curcumin, DMC, BDMC) plasmatic concentrations | from 0 to 8 hours
  AUC of curcuminoids separately (curcumin, DMC, BDMC) plasmatic concentrations from 0 to 8 hours (AUC0-8h, expressed in µg.h/mL);
AUC of curcuminoids metabolites plasmatic concentrations | from 0 to 8 hours
  AUC of curcuminoids metabolites plasmatic concentrations from 0 to 8 hours (AUC0-8h, expressed in µg.h/mL);
AUC of total curcuminoids plasmatic concentration normalized to curcuminoids intake | from 0 to infinity
  AUC of total curcuminoids plasmatic concentration from 0 to infinity normalized to curcuminoids intake (AUC0-infinity/dose, expressed in µg.h/mL/mg);
AUC of total curcuminoids plasmatic concentration | from 0 to infinity
  AUC of total curcuminoids plasmatic concentration from 0 to infinity (AUC0-infinity, expressed in µg.h/mL);
AUC of curcuminoids separately (curcumin, DMC, BDMC) plasmatic concentrations | from 0 to infinity
  AUC of curcuminoids separately (curcumin, DMC, BDMC) plasmatic concentrations from 0 to infinity (AUC0-infinity, expressed in µg.h/mL);
AUC of curcuminoids metabolites plasmatic concentrations | from 0 to infinity
  AUC of curcuminoidsmetabolites plasmatic concentrations from 0 to infinity (AUC0-infinity, expressed in µg.h/mL);
Peak of total curcuminoids plasmatic concentration normalized to curcuminoids intake | 24hours
  Peak of total curcuminoids plasmatic concentration normalized to curcuminoids intake (Cmax/dose, expressed in µg/mL/mg);
Peak of total curcuminoids plasmatic concentration | 24hours
  Peak of total curcuminoids plasmatic concentration (Cmax, expressed in µg/mL);
Peak of curcuminoids separately plasmatic concentrations | 24hours
  Peak of curcuminoids separately plasmatic concentrations (Cmax, expressed in µg/mL);
Peak of curcuminoids metabolites plasmatic concentrations | 24hours
  Peak of curcuminoids metabolites plasmatic concentrations (Cmax, expressed in µg/mL);
Half-life of total curcuminoids in plasma | 24hours
  Half-life of total curcuminoids in plasma (t1/2, expressed in minutes);
Half-life of curcuminoids separately (curcumin, DMC, BDMC) in plasma | 24hours
  Half-life of curcuminoids separately (curcumin, DMC, BDMC) in plasma (t1/2, expressed in minutes);
Half-life of curcuminoids metabolites in plasma | 24hours
  Half-life of curcuminoids metabolites in plasma (t1/2, expressed in minutes);
Terminal elimination rate constant of total curcuminoids in plasma (λz) | 24hours
  Terminal elimination rate constant of total curcuminoids in plasma (λz);
Terminal elimination rate constant curcuminoids separately (curcumin, DMC, BDMC) in plasma (λz) | 24hours
  Terminal elimination rate constant curcuminoids separately (curcumin, DMC, BDMC) in plasma (λz);
Terminal elimination rate constant curcuminoids metabolites in plasma (λz) | 24hours
  Terminal elimination rate constant curcuminoids metabolites in plasma (λz);
Time to peak of total curcuminoids plasmatic concentrations | 24hours
  Time to peak of total curcuminoids plasmatic concentration in plasma (Tmax, expressed in minutes)
Time to peak of curcuminoids separately (curcumin, DMC, BDMC) plasmatic concentrations | 24hours
  Time to peak of plasmatic concentrations curcuminoids separately (curcumin, DMC, BDMC) in plasma (Tmax, expressed in minutes);
Time to peak of curcuminoids metabolites plasmatic concentrations | 24hours
  Time to peak of plasmatic concentrations curcuminoids metabolites in plasma (Tmax, expressed in minutes);
Relative bioavailability | from 0 to 24 hours
  Relative bioavailability from 0 to 24 hours defined as the ratio of dose-normalized AUC0-24h of total curcuminoids for the different tested formulation to the dose-normalized AUC0-24h obtained for the reference product (turmeric extract 95% curcuminoids).

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Fança-Berthon, PhD, Study Director — Naturex
Locations (1):
- Biofortis Mérieux NutriSciences, Saint-Herblain, France

REFERENCES:
- [Derived] Fanca-Berthon P, Tenon M, Bouter-Banon SL, Manfre A, Maudet C, Dion A, Chevallier H, Laval J, van Breemen RB. Pharmacokinetics of a Single Dose of Turmeric Curcuminoids Depends on Formulation: Results of a Human Crossover Study. J Nutr. 2021 Jul 1;151(7):1802-1816. doi: 10.1093/jn/nxab087. PMID 33877323